CLINICAL TRIAL: NCT01443598
Title: Observational Study of Patients With Pre Capillary Pulmonary Hypertension
Brief Title: Pulmonary Hypertension in Interstitial Lung Disease
Acronym: HYPID
Status: Completed | Type: Observational
Sponsor: Groupe d'Etudes et de Recherche sur les Maladies Orphelines Pulmonaires (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Vincent COTTIN, Professor V. Cottin, Groupe d'Etudes et de Recherche sur les Maladies Orphelines Pulmonaires
Other Study IDs: GERMOP-002
Record Dates: First submitted 2011-09-28; First posted 2011-09-29 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Pulmonary Arterial Hypertension; Diffuse Interstitial Lung Disease
Keywords: Pulmonary arterial hypertension,; Interstitial lung disease at HRCT
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum and plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
HYPID study is an observational and prospective study of patients with interstitial lung disease and pre capillary hypertension diagnosed by right heart sided catheterization. The primary aim of the study is to identify prognostic factors.

DETAILED DESCRIPTION:
Pre capillary pulmonary hypertension (PH) may be present in patients with diffuse interstitial lung disease.

In this context, PH represents an important factor of morbidity and mortality for these patients.

One of the purposes of HYPID is to determine predictive factors of mortality within this cohort of patients.

In order to reach that aim,the study includes an evaluation based on exams conducted for the routine follow-up of patients. Each patient will be followed during 2 years at least.

ELIGIBILITY:
Inclusion Criteria:

* pre capillary pulmonary hypertension at right heart sided catheterization with: mPAP > or = 25 mmHg,PCWP < or = 15 mmHg
* interstitial lung disease with diffuse infiltrative opacities on chest CT scan

Exclusion Criteria:

* pulmonary hypertension related to a thromboembolic disease
* respiratory disease other than diffuse interstitial lung disease
* any etiological factor of pulmonary arterial hypertension based on DANA POINT classification other than diffuse interstitial lung disease
* any progressive disease associated to a life expectancy less than 6 months other than pulmonary hypertension, diffuse interstitial lung disease and respiratory insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pre capillary pulmonary hypertension and interstitial lung disease at HRCT
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2 years
  Determine predictive factors of mortality

SECONDARY OUTCOMES:
Progression-free survival (1) | 2 years
  Determine cause of death
Progression-free survival (2) | 2 years
  Determine survival and time to worsening
Progression-free survival (3) | 2 years
  Analyse clinical, functional respiratory, hemodynamic features and changing characteristics of pulmonary hypertension
Progression-free survival (4) | 2 years
  Document the efficacy of PH specific treatment
Progression-free survival (5) | 2 years
  Evaluate the level of pulmonary arterial hypertension and compare the functional characteristics of patients with moderate or severe pulmonary hypertension
Progression-free survival (6) | 2 years
  Analyse clinical, functional respiratory, hemodynamic features and changing characteristics of pulmonary hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Cottin, MD, Principal Investigator — Hospices Civils de Lyon / University Lyon I
Locations (1):
- Louis Pradel Hospital (Bâtiment A4), Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: website National French Reference Center for rare lung diseases — http://maladies-pulmonaires-rares.fr/